CLINICAL TRIAL: NCT00682539
Title: A Randomized, Double-masked Study With Intraocular Anti-VEGF (Avastin®/Lucentis®) Compared With Intraocular Triamcinolone (Volon A®) in Patients With Clinical Significant Diabetic Macular Edema
Brief Title: Intraocular Anti-VEGF Compared With Intraocular Triamcinolone in Patients With Diabetic Macular Edema
Acronym: TRIASTIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Katharina Kriechbaum, Ass.Prof.Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRIASTIN Study
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic retinopathy; macular edema; intravitreal Avastin/ Triamcinolone / Lucentis
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema | interventions — Bevacizumab; Triamcinolone; salicylhydroxamic acid; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Avastin (Active Comparator): 15 patients with clinical significant macular edema receive an injection of 2,5 mg Avastin every month. After three initial injections of Avastin re-injection is performed if the central retinal thickness measured with optical coherence tomography (Stratus OCT, Zeiss) stays more than 300 microns. If the Central retinal thickness decreases under 300 microns a sham injection is performed.
  Interventions: Drug: Bevacizumab (Avastin); Drug: Sham
- Triamciolone (Active Comparator): 30 patients with a clinical significant diabetic macular edema receive an intraocular injection of 8mg triamcinolone at baseline under sterile conditions. 1 and 2 month after the baseline injection, patients receive a sham injection. After three month re-injection of 8mg Triamcinolone is performed if the central retinal thickness measured with optical coherence tomography (Stratus OCT, Zeiss) stays more than 300 microns. If the Central retinal thickness decreases under 300 microns patients will receive a sham injection. In between two injection of 8mg Triamcinolone must be an temporal interval of at least 3 months.
  Interventions: Drug: Triamcinolone; Drug: Sham
- Lucentis (Active Comparator): 15 patients with clinical significant macular edema receive an injection of 0,5 mg Lucentis every month. After three initial injections of Lucentis re-injection is performed if the central retinal thickness measured with optical coherence tomography (Stratus OCT, Zeiss) stays more than 300 microns. If the Central retinal thickness decreases under 300 microns a sham injection is performed.
  Interventions: Procedure: Lucentis

INTERVENTIONS:
Drug: Bevacizumab (Avastin) — The intravitreal injection of Bevacizumab (Avastin®) is performed in the operating room under sterile conditions. The patient receives an initial drop of lidocaine 4% into the study eye followed by betaisodona solution. Then the lid margins, the lids and the periocular skin are washed carefully with betaisodona. The eye is draped in a sterile fashion. A sterile lid speculum is inserted by the surgeon. Another drop of betaisodona is applied into the eye. A circle is used to mark the injection site 3.5mm from the limbus in the inferior temporal quadrant. The injection is given at the marked site, slowly, at a 90 degree angle. After injecting the total volume of 0.1ml the needle is slowly withdrawn. Another drop of betaisodona is given as well as an antibiotic/steroid ointment.
  Other Names: Avastin
  Arms: Avastin
Drug: Triamcinolone — The intravitreal injection of triamcinolone (Volon A®) is performed in the operating room under sterile conditions at baseline. The patient receives an initial drop of lidocaine 4% into the study eye followed by betaisodona solution. Then the lid margins, the lids and the periocular skin are washed carefully with betaisodona. The eye is draped in a sterile fashion. A sterile lid speculum is inserted by the surgeon. Another drop of betaisodona is applied into the eye. A circle is used to mark the injection site 3.5mm from the limbus in the inferior temporal quadrant. The injection is given at the marked site, slowly, at a 90 degree angle. After injecting the total volume of 0.1ml the needle is slowly withdrawn. Another drop of betaisodona is given as well as an antibiotic/steroid ointment.
  Other Names: Volon A
  Arms: Triamciolone
Drug: Sham — Patients receiving sham intravitreal injections do not receive an actual injection of study drug. The injecting physician performing the sham injection will be unmasked to the treatment to the treatment assignment regarding active versus sham. The injecting physician will perform the same pre-injection procedures for the patients receiving bevacizumab or triamcinolone, An empty syringe without a needle will be used in the sham injection. The injecting physician will mimic an intraocular injection by making contact with the conjunctiva and applying pressure without the needle. Immediately following the sham injection, the injecting physician will perform the same post-injection procedures as those performed on patients receiving bevacizumab or triamcinolone.
  Other Names: sham injection
  Arms: Avastin; Triamciolone
Procedure: Lucentis — The intravitreal injection of Ranibizumab (Lucentis®) is performed in the operating room under sterile conditions. The patient receives an initial drop of lidocaine 4% into the study eye followed by betaisodona solution. Then the lid margins, the lids and the periocular skin are washed carefully with betaisodona. The eye is draped in a sterile fashion. A sterile lid speculum is inserted by the surgeon. Another drop of betaisodona is applied into the eye. A circle is used to mark the injection site 3.5mm from the limbus in the inferior temporal quadrant. The injection is given at the marked site, slowly, at a 90 degree angle. After injecting the total volume of 0.05ml the needle is slowly withdrawn. Another drop of betaisodona is given as well as an antibiotic/steroid ointment.
  Arms: Lucentis

SUMMARY:
The purpose of this study is to investigate the change in macular edema and the absolute change in visual acuity following intravitreal administered injections of Bevacizumab (Avastin®) or Ranibizumab (Lucentis®) compared with Triamcinolone (Volon A®) in patients with clinical significant diabetic macular edema.

The investigators monitor the change in macular edema measured with standard optical coherence tomography (OCT) and the absolute change in visual acuity analyzed by standardized charts according to the protocol used in the Early Retreatment in Diabetic Retinopathy Study (ETDRS).

DETAILED DESCRIPTION:
Diabetes mellitus is the most common endocrine disease in developed countries, with prevalence estimates ranging between 2 to 5% of the world's population. Diabetic retinopathy and diabetic macular edema are common microvascular complications in diabetic patients and may lead to decreasing of visual acuity, eventually to blindness. The Wisconsin Epidemiologic Study found an incidence of macular edema of 20.1% in the younger-onset group and of 14 to 25% in patients with type 2 diabetes mellitus over a period of 10 years.

Diabetic macular edema is characterized by the accumulation of extracellular fluid in Henle´s layer and the inner nuclear layer of the retina. There pathogenesis involves the interaction of several factors: the breakdown of the blood-retinal-barriers, production of biochemical factors, tissue hypoxia, retinal circulatory changes and vitreous tractions.

Laser photocoagulation is the most common treatment modality for diabetic macular edema. Perifoveal focal/grid laser coagulation was found to be effective saving the visual acuity in only 50% of patients with diabetic macular edema and just 3-14% of treated patients had an improved visual acuity post-operatively. The decent results of laser coagulation are associated with potential side effects as paracentral scotomas[4], change of color discrimination, development of epiretinal gliosis and subretinal fibrosis and expansion of laser scar size.

In the past few years, several studies investigating the effect of intravitreal steroids such as triamcinolone in patients with diabetic macular edema found a significant reduction in macular edema. Therefore intravitreal steroids have become part of standard therapy in the treatment of diabetic macular edema.

Furthermore, some studies showed that the vascular endothelial growth factor (VEGF) is the major angiogenic stimulus responsible for increase of vasopermeability, cell proliferation and angiogenesis in diabetic retinopathy (DRP). Evaluation of VEGF levels in the vitreous have indicated a role for VEGF in diabetic macular edema: vitreous samples of patients with diabetic macular edema contain elevated VEGF concentration and injection of VEGF in experimental studies led to breakdown of the blood-retina barrier.

Not only in age-related macular degeneration but also in other diseases like in diabetic macular edema we can find an increasing evidence for a therapeutic role of anti-VEGF drugs. Intravitreal injections have become the most favored treatment procedure for administering anti-VEGF drugs.

The side effects and the modest results of laser treatment on the visual acuity in diabetic macular edema led to studies using anti-VEGF therapy. Unpublished study results on the aptamer pegaptanib (Macugen®) are promising. A study using the antibody fragment Ranibizumab (Lucentis®) is in progress.

Currently there is one anti-VEGF drug already on the market: Bevacizumab (Avastin®), which has approved as intravenous infusion for the treatment of metastatic colo-rectal cancer. Previous studies have shown that systemic use of Bevacizumab (Avastin®) can obtain very promising results on patients with choroidal neovascularisation (CNV) by age-related macular degeneration. This drug, a monoclonal full-length antibody, designed to bind all isoforms of VEGF, is a large molecule. But case reports in patients with CNV caused by age-related macular degeneration and with macular edema from central retinal vein occlusion indicate that intravitreally given Bevacizumab (Avastin™) is effective in diseases originating from the choroids and also the retina. These findings imply a sufficient penetration of the retina by Bevacizumab (Avastin®).

A recent study investigating the effect of intravitreal bevacizumab (Avastin®) in patients with diabetic macular edema found a significant reduction in macular edema.

Based on these new findings and the important role of VEGF in diabetic macular edema and in proliferative diabetic retinopathy, we propose a double-masked, randomised pilot study for treatment of diabetic macular edema with intravitreally administered anti VEGF (Avastin®/Lucentis®) compared with intravitreally administered triamcinolone (VolonA®).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients with type 1 or type 2 diabetes mellitus
* Patients with diabetic macular edema with center involvement
* Central macular thickness (macular edema) of at least 300 microns in the central subfield as measured by OCT
* Best corrected visual acuity, using ETDRS charts, of 20/25 to 20/400 (Snellen equivalent) in the study eye
* Patients with decrease in vision in the study eye due to foveal thickening from diabetic macular edema and not to other causes, in the opinion of the investigator
* Patients without a necessity for panretinal laser photocoagulation for at least 3 months after study inclusion
* If both eyes are eligible, the one with the worse visual acuity will be selected for study treatment unless, based on medical reason, the investigator deems the other eye have got more benefit from study treatment. The other eye will be treated with Grid laser coagulation.

Exclusion Criteria:

* A condition that would preclude a patient for participation in the study in opinion of investigator, e.g., unstable medical status including glycemic control and blood pressure
* History of systemic corticosteroids within 3 months prior to randomization or topical, rectal or inhaled corticosteroids in current use more than 3 times per week

Prior/Concomitant Treatment

* Macular laser photocoagulation
* Panretinal laser photocoagulation within the past 3 months
* Previous treatment with intravitreal or sub-Tenon triamcinolone within the past 3 months in the study eye
* Previous participation in clinical trial involving anti-angiogenic drugs (pegaptanib sodium, ranibizumab, anecortave acetate, protein kinase C inhibitor, etc.)
* History of submacular surgery or other surgical intervention for diabetic macular edema in the study eye Diabetic Retinopathy Characteristics
* High risk proliferative diabetic retinopathy in the study eye without complete panretinal laser photocoagulation and having a risk for intravitreal bleeding Concurrent Ocular Conditions
* Active intraocular inflammation (grade trace or above) in either eye
* Vitreomacular traction in the study eye evident by OCT
* Ocular disorders in the study eye including retinal vascular occlusion, retinal detachment, macular hole, choroidal neovascularisation
* Intraocular surgery (including cataract surgery, YAG laser capsulotomy) in the study eye within 3 months preceding Day 0
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥25 mmHg despite treatment with anti-glaucoma medication)
* History of glaucoma filtration surgery, corneal transplantation in the study eye Concurrent Systemic Conditions
* History of myocardial infarction (in anamnesis or signs in ECG)
* History of congestive heart failure
* History of stroke or transient ischemic attacks
* Significant abnormalities on laboratory testing (signs on failure of kidney, liver disease)
* Premenopausal women not using adequate contraception and pregnant or nursing women
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications
* Current treatment for active systemic infection Other
* History of allergy to fluorescein, not amenable to treatment
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality to be analyzed and graded
* Inability to comply with study or follow up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Schmidt-Erfurth, MD, Study Chair — Medical University of Vienna, Dept. of Ophthalmology; Georg Rainer, MD, Principal Investigator — Medical University of Vienna, Dept. of Ophthalmology
Locations (1):
- Dept. of Ophthalmology, Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rittiphairoj T, Mir TA, Li T, Virgili G. Intravitreal steroids for macular edema in diabetes. Cochrane Database Syst Rev. 2020 Nov 17;11(11):CD005656. doi: 10.1002/14651858.CD005656.pub3. PMID 33206392
- [Derived] Karst SG, Lammer J, Mitsch C, Schober M, Mehta J, Scholda C, Kundi M, Kriechbaum K, Schmidt-Erfurth U. Detailed analysis of retinal morphology in patients with diabetic macular edema (DME) randomized to ranibizumab or triamcinolone treatment. Graefes Arch Clin Exp Ophthalmol. 2018 Jan;256(1):49-58. doi: 10.1007/s00417-017-3828-1. Epub 2017 Oct 28. PMID 29080915

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study patients were recruited between 2007 and 2014 at the outpatient clinic of the Department of Ophthalmology, Medical University Vienna, Austria.
Groups:
- Avastin: 15 patients with clinical significant macular edema receive an injection of 2,5 mg Avastin every month. After three initial injections of Avastin re-injection is performed following a predefined protocol.
- Triamciolone: 30 patients with a clinical significant diabetic macular edema receive an intraocular injection of 8mg triamcinolone at baseline under sterile conditions. 1 and 2 month after the baseline injection, patients receive a sham injection. After three month re-injection of 8mg Triamcinolone is performed as needed following a predefined protocol. In between two injection of 8mg Triamcinolone must be an temporal interval of at least 3 months.
- Lucentis: 15 patients with clinical significant macular edema receive an injection of 0,5 mg Lucentis every month. After three initial injections of Lucentis re-injection is performed as needed following a predefined protocol.
Period: Bevacizumab vs Triamcinolone
Arm/Group | Avastin | Triamciolone | Lucentis
Started | 18 | 16 | 0
Completed | 15 | 15 | 0
Not Completed | 3 | 1 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0
Period: Ranibizumab vs Triamcinolone
Arm/Group | Avastin | Triamciolone | Lucentis
Started | 0 (Two independent periods.) | 18 (None of the patients of the 1st period was included in the second period.) | 18 (Both periods recruited independently following the same criteria.)
Completed | 0 | 15 | 10
Not Completed | 0 | 3 | 8
Not completed — Lost to Follow-up | 0 | 3 | 8

BASELINE CHARACTERISTICS:
Population: The sample size will be calculated so that a true group difference in changes of macular edema of 50 μm can be detected with a probability of 90 %. Repeated-measures-ANOVA will be used to reveal differences between macular edema measurements before and after treatment and between groups
Groups:
- Avastin: After a loading dose of three monthly injections of 2.5mg Avastin, PRN treatment based on predefined morphological and functional retreatment criteria, that were reassessed monthly.
- Triamciolone: Baseline injection of 8mg intravitreally applied triamcinolone was followed by two sham injections at month 1 and 2. Sham injections were only mimicked without penetration of the ocular globe after the same pre-injection procedure. Beginning at month 3 patients were treated as needed (PRN) based on predefined morphological and functional retreatment criteria, that were reassessed monthly. Triamcinolone was injected no more than every three months intermitted by sham injections to maintain patient masking.
- Lucentis: After a loading dose of three monthly injections of 0.5mg Lucentis, PRN treatment based on predefined morphological and functional retreatment criteria, that were reassessed monthly.
- Total: Total of all reporting groups
Arm/Group | Avastin | Triamciolone | Lucentis | Total
Number analyzed (Participants) | 15 | 30 | 10 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 19 | 6 | 36
  >=65 years | 4 | 11 | 4 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 14 | 2 | 20
  Male | 11 | 16 | 8 | 35

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of the Treatment Assessed With Visual Acuity Measured by ETDRS Charts.
Description: Efficacy of the treatment with intravitreal administered injections of anti VEGF (Bevacizumab (Avastin®) or Ranibizumab (Lucentis®) ) compared with triamcinolone (Volon A®) in patients with diabetic macular edema is examined using Visual acuity measurements with ETDRS charts: units: logMAR; scale range: -0.1 to 1.0; higher values are considered worse outcome
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Avastin: Loading dose of three monthly 2.5mg Avastin injections followed by PRN treatment.
- Triamciolone: Initial 8mg intravitreally applied Triamcinolone followed by two sham injections. PRN treatment from month 3.
- Lucentis: Loading dose of three monthly 0.5mg Lucentis injections followed by PRN treatment.
Arm/Group | Avastin | Triamciolone | Lucentis
Number analyzed (Participants) | 15 | 30 | 10
logMAR | 0.18 (0.12) | 0.36 (0.19) | 0.18 (0.15)

2. Primary Outcome: Efficacy of the Treatment Assessed by Standard Optical Coherence Tomography (OCT)
Description: Efficacy of the treatment with intravitreal administered injections of anti VEGF (Bevacizumab (Avastin®) or Ranibizumab (Lucentis®) ) compared with triamcinolone (Volon A®) in patients with diabetic macular edema is measured with standard Optical Coherence Tomography - (OCT): units: µm; scale range: 200-800; higher values are considered worse outcome
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Avastin | Triamciolone | Lucentis
Number analyzed (Participants) | 15 | 30 | 10
µm | 351 (93) | 357 (152) | 389 (137)

3. Secondary Outcome: To Explore the Structural Mechanisms of the Effect on Diabetic Macular Edema as Assessed by Fluorescein Angiography and Ultra High-resolution Optical Coherence Tomography. To Observe the Changes in Retinal Function a Microperimetry is Assessed.
Description: Area of leakage and non perfusion is measured in FA, morphologic details like presence of cysts or sub retinal fluid is evaluated in OCT. Data is still under evaluation.
Time Frame: 12 month
Reporting Status: Not Posted, anticipated posting 2016-06

ADVERSE EVENTS:
Groups:
- Avastin: Patients with clinical significant macular edema receive an injection of 2,5 mg Avastin every month. After three initial injections of Avastin re-injection is performed as needed.
- Triamciolone: 30 patients with a clinical significant diabetic macular edema receive an intraocular injection of 8mg triamcinolone at baseline under sterile conditions. 1 and 2 month after the baseline injection, patients receive a sham injection. After three month re-injection of 8mg Triamcinolone is performed if needed. In between two injection of 8mg Triamcinolone must be an temporal interval of at least 3 months.
- Lucentis: 15 patients with clinical significant macular edema receive an injection of 0,5 mg Lucentis every month. After three initial injections of Lucentis re-injection is performed if needed.
Arm/Group | Avastin | Triamciolone | Lucentis
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/30 | 0/10
Other Adverse Events (participants affected / at risk) | 0/15 | 7/30 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin (N=15) | Triamciolone (N=30) | Lucentis (N=10)
IOP elevation >25mmHg (Eye disorders) | 0 | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes